CLINICAL TRIAL: NCT00653887
Title: Modifications of the Anal Muscle Cortical Excitability Area After Biofeedback Training
Brief Title: Biofeedback and Cortical Excitability
Acronym: Biofeedback
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Procedure needs to be changed
Sponsor: University Hospital, Rouen (Other)
Collaborators: Coloplast A/S (Industry)
Responsible Party: Leroi, Physiology unit
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 2007/054/HP; 2007- A00652-51
Record Dates: First submitted 2008-04-02; First posted 2008-04-07 (Estimated); Last update posted 2012-02-16 (Estimated); Status verified 2012-02

CONDITIONS: Incontinence; Constipation
Keywords: Biofeedback; anal sphincter; cortical excitability; magnetic stimulation; incontinence; constipation
MeSH Terms: conditions — Constipation | interventions — Biofeedback, Psychology

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): biofeedback (active group)
  Interventions: Other: Biofeedback
- B (Placebo Comparator): discussion about digestive tract (placebo group)
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Biofeedback — 4 sessions of biofeedback one session each week
  Arms: A
Other: Placebo — 4 sessions, one each week, of discussion about anorectal disease
  Arms: B

SUMMARY:
Looking for a modification of the cortical excitability of the motor area corresponding to the external anal sphincter after biofeedback sessions.

DETAILED DESCRIPTION:
Introduction: Nervous control of pelvic floor is not much known. The dysfunction of this musculature, and particularly of the external anal sphincter, is a frequent cause of anal incontinence and/or dyschesia. Biofeedback training is often offered to patients suffering from incontinence or constipation. However, its mechanisms of action is still controversial.

Objective of the study: to compare excitability of the cortical area responsible for control volunteer of the external anal sphincter in healthy subjects before and after 4 biofeedback sessions.

Subjects and methodology: we offer to perform two groups of 12 healthy subjects (one active and one control group) without any neurological or digestive disease and having never performed biofeedback. In each group, cortical excitability will be evaluated by cortical magnetic stimulation (curve intensity/amplitude, silent period, inter-stimulus period, motor threshold) before and after 4 biofeedback sessions (one session by week) in active group or 4 placebo sessions (placebo group).

We hope to show a modification of cortical excitability in subjects performing biofeedback compared to others.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers between 18 years old and 35 years old
* Right handed*

Exclusion Criteria:

* Pregnancy
* Pace-maker or other metallic piece implanted in the body
* Neurological disease
* Epilepsy
* Digestive disease
* Traumatic delivery
* Anorectal surgery
* Biofeedback
* Psychiatric disease
* Treatment anti-epileptic, hypnotic, psychotropic
* Participation to a previous protocol within 1 month

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2008-01; Primary Completion 2009-09 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
external anal sphincter motor threshold silent period double-pulse stimulation: inter-stimulus interval amplitude and duration of external anal sphincter contraction | final

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Marie LEROI, PhD, Principal Investigator — CHU Rouen
Locations (1):
- Physiology Unit - Rouen university Hospital, Rouen, France